CLINICAL TRIAL: NCT01859988
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study Investigating the Efficacy, Safety, Pharmacokinetic and Biomarker Profiles of Dupilumab (REGN668) Administered to Adult Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Study of Dupilumab Administered to Adult Patients With Moderate-to-Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R668-AD-1021
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Atopic Dermatitis
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo qw (Experimental): Two subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1 followed by a single injection every week (qw) from Week 1 to Week 15.
  Interventions: Drug: Placebo
- Dupilumab 300 mg qw (Experimental): Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection qw from Week 1 to Week 15.
  Interventions: Drug: Dupilumab
- Dupilumab 300 mg q2w (Experimental): Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single injection of Placebo (for Dupilumab) alternating with single 300 mg injection of Dupilumab every 2 weeks (q2w) from Week 1 to Week 15.
  Interventions: Drug: Dupilumab; Drug: Placebo
- Dupilumab 200 mg q2w (Experimental): Two subcutaneous injections of Dupilumab 200 mg (for a total of 400 mg) as a loading dose on Day 1, followed by a single injection of Placebo (for Dupilumab) alternating with single 200 mg injection of Dupilumab q2w from Week 1 to Week 15.
  Interventions: Drug: Dupilumab; Drug: Placebo
- Dupilumab 300 mg q4w (Experimental): Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection of Dupilumab every 4 weeks (q4w) and Placebo (for Dupilumab) qw when Dupilumab not administered from Week 1 to Week 15.
  Interventions: Drug: Dupilumab; Drug: Placebo
- Dupilumab 100 mg q4w (Experimental): Two subcutaneous injections of Dupilumab 200 mg (for a total of 400 mg) as a loading dose on Day 1, followed by a single 100 mg injection of Dupilumab q4w and Placebo (for Dupilumab) qw when Dupilumab not administered from Week 1 to Week 15.
  Interventions: Drug: Dupilumab; Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab
  Other Names: REGN668; SAR231893; Dupixent
  Arms: Dupilumab 100 mg q4w; Dupilumab 200 mg q2w; Dupilumab 300 mg q2w; Dupilumab 300 mg q4w; Dupilumab 300 mg qw
Drug: Placebo
  Arms: Dupilumab 100 mg q4w; Dupilumab 200 mg q2w; Dupilumab 300 mg q2w; Dupilumab 300 mg q4w; Placebo qw

SUMMARY:
To assess the efficacy of multiple dupilumab dose-regimens, compared to placebo, in adult participants with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
The inclusion criteria included, but were not limited to, the following:

1. Chronic Atopic Dermatitis that had been present for at least 3 years
2. History of inadequate response to out-patient treatment with topical medications, or for whom topical treatments were otherwise inadvisable (e.g, because of important side effects or safety risks)
3. Willing and able to comply with all clinic visits and study-related procedures

The exclusion criteria included, but were not limited to, the following:

1. Prior treatment with dupilumab (REGN668/SAR231893)
2. Presence of certain laboratory abnormalities at the screening visit
3. Treatment with an investigational drug within 8 weeks of baseline visit
4. Treatment with a live (attenuated) vaccine within 12 weeks before the baseline visit
5. Certain other treatments and medical procedures undertaken within a particular time frame prior to the baseline visit
6. Known history of human immunodeficiency virus (HIV) infection
7. History of malignancy within 5 years before the baseline visit (with certain exceptions)
8. Planned surgical procedure during the length of the study
9. High risk of parasite infection
10. Any other medical or psychological condition that in the opinion of the investigator or the sponsor's medical monitor, would place the participants at risk, interfere with participation in the study or interfere with interpretation of study results
11. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (84):
- United States (25):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Tucson, Arizona
  - Bakersfield, California
  - San Diego, California
  - Santa Monica, California
  - Jacksonville, Florida
  - Ormond Beach, Florida
  - Skokie, Illinois
  - New Orleans, Louisiana
  - Andover, Massachusetts
  - Boston, Massachusetts
  - Troy, Michigan
  - St Louis, Missouri
  - New York, New York
  - Rochester, New York
  - Winston-Salem, North Carolina
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Johnston, Rhode Island
  - Greer, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Seattle, Washington
- Canada (12):
  - Vancouver (2 Locations), British Columbia
  - Winnipeg, Manitoba
  - Barrie, Ontario
  - Hamilton, Ontario
  - Markham, Ontario
  - Oakville, Ontario
  - Peterborough, Ontario
  - Richmond Hill, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
  - Saint-Hyacinthe, Quebec
  - Québec
- Czechia (5):
  - Kutná Hora
  - Náchod
  - Prague
  - Svitavy
  - Ústí nad Labem
- Germany (17):
  - Augsburg
  - Baden
  - Berlin
  - Bonn
  - Dresden
  - Dülmen
  - Frankfurt am Main
  - Frankfurt/Main, Hessen
  - Gera
  - Hamburg
  - Heidelberg
  - Kiel
  - Mahlow
  - Munich
  - Münster
  - Osnabrück
  - Tübingen
- Hungary (6):
  - Borsod-Abauj-Zemplen
  - Budapest
  - Kaposvár
  - Szeged
  - Szolnok
  - Tolna
- Japan (12):
  - Fukuoka
  - Hokkaido
  - Saitama
  - Tokyo, Bunkyo-ku
  - Tokyo, Chiyoda-ku
  - Tokyo, Nakano-ku
  - Tokyo, Nerima-ku
  - Tokyo, Shibuya-ku
  - Tokyo, Shinagawa-ku
  - Tokyo, Shinjuku-ku (2 Locations)
  - Tokyo, Suginami-ku (2 Locations)
  - Yokohama
- Poland (7):
  - Gdansk (2 Locations)
  - Katowice
  - Lodz
  - Lublin
  - Poznan
  - Warsaw (2 Locations)
  - Wroclaw

REFERENCES:
- [Result] Thaci D, Simpson EL, Beck LA, Bieber T, Blauvelt A, Papp K, Soong W, Worm M, Szepietowski JC, Sofen H, Kawashima M, Wu R, Weinstein SP, Graham NM, Pirozzi G, Teper A, Sutherland ER, Mastey V, Stahl N, Yancopoulos GD, Ardeleanu M. Efficacy and safety of dupilumab in adults with moderate-to-severe atopic dermatitis inadequately controlled by topical treatments: a randomised, placebo-controlled, dose-ranging phase 2b trial. Lancet. 2016 Jan 2;387(10013):40-52. doi: 10.1016/S0140-6736(15)00388-8. Epub 2015 Oct 8. PMID 26454361
- [Result] Simpson EL, Bieber T, Eckert L, Wu R, Ardeleanu M, Graham NM, Pirozzi G, Mastey V. Patient burden of moderate to severe atopic dermatitis (AD): Insights from a phase 2b clinical trial of dupilumab in adults. J Am Acad Dermatol. 2016 Mar;74(3):491-8. doi: 10.1016/j.jaad.2015.10.043. Epub 2016 Jan 14. PMID 26777100
- [Result] Simpson EL, Gadkari A, Worm M, Soong W, Blauvelt A, Eckert L, Wu R, Ardeleanu M, Graham NMH, Pirozzi G, Sutherland ER, Mastey V. Dupilumab therapy provides clinically meaningful improvement in patient-reported outcomes (PROs): A phase IIb, randomized, placebo-controlled, clinical trial in adult patients with moderate to severe atopic dermatitis (AD). J Am Acad Dermatol. 2016 Sep;75(3):506-515. doi: 10.1016/j.jaad.2016.04.054. Epub 2016 Jun 4. PMID 27268421
- [Derived] Paller AS, Silverberg JI, Cork MJ, Guttman-Yassky E, Lockshin B, Irvine AD, Kim MB, Kabashima K, Chen Z, Lu Y, Bansal A, Rossi AB, Shabbir A. Efficacy and Safety of Dupilumab in Patients With Erythrodermic Atopic Dermatitis: A Post Hoc Analysis of 6 Randomized Clinical Trials. JAMA Dermatol. 2023 Mar 1;159(3):255-266. doi: 10.1001/jamadermatol.2022.6192. PMID 36723913
- [Derived] Kamal MA, Davis JD, Kovalenko P, Srinivasan K, Simpson EL, Nakahara T, Sugaya M, Igarashi A, Ardeleanu M, Xu C, Arima K. Pharmacokinetics, pharmacodynamics, and exposure-efficacy of dupilumab in adults with atopic dermatitis. Clin Transl Sci. 2022 Oct;15(10):2342-2354. doi: 10.1111/cts.13363. Epub 2022 Aug 20. PMID 35986664
- [Derived] Silverberg JI, Simpson EL, Guttman-Yassky E, Cork MJ, de Bruin-Weller M, Yosipovitch G, Eckert L, Chen Z, Ardeleanu M, Shumel B, Hultsch T, Rossi AB, Hamilton JD, Orengo JM, Ruddy M, Graham NMH, Pirozzi G, Gadkari A. Dupilumab Significantly Modulates Pain and Discomfort in Patients With Atopic Dermatitis: A Post Hoc Analysis of 5 Randomized Clinical Trials. Dermatitis. 2021 Oct 1;32(1S):S81-S91. doi: 10.1097/DER.0000000000000698. PMID 33165005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 95 study sites in 7 countries. A total of 452 participants were screened between 15 May 2013 and 10 January 2014. 380 participants were randomized and 379 were treated. 72 participants were screen failures mainly due to exclusion criteria met and inclusion criteria not met.
Pre-assignment Details: Randomization was stratified by disease severity (moderate Investigator's global assessment [IGA] = 3 versus severe IGA = 4 atopic dermatitis) and region (Japan versus rest of world). Assignment to arms was done centrally in 1:1:1:1:1:1 ratio for Dupilumab (300 mg qw; 300 mg q2w; 200 mg q2w; 300 mg q4w and 100 mg q4w) and Placebo.
Groups:
- Dupilumab 300 mg qw: Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection every week (qw) from Week 1 to Week 15.
- Dupilumab 300 mg q4w: Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection of Dupilumab every 4 weeks (q4w) and Placebo (for Dupilumab) qw (when Dupilumab not administered) from Week 1 to Week 15.
- Dupilumab 100 mg q4w: Two subcutaneous injections of Dupilumab 200 mg (for a total of 400 mg) as a loading dose on Day 1, followed by a single 100 mg injection of Dupilumab q4w and Placebo (for Dupilumab) qw (when Dupilumab not administered) from Week 1 to Week 15.
- Placebo: Two subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1 followed by a single injection qw from Week 1 to Week 15.
Period: Overall Study
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Started | 63 | 64 | 62 | 65 | 65 | 61
Treated | 63 | 64 | 61 | 65 | 65 | 61
Completed | 52 | 52 | 34 | 55 | 42 | 42
Not Completed | 11 | 12 | 28 | 10 | 23 | 19
Not completed — Withdrawal by Subject | 6 | 3 | 4 | 3 | 2 | 2
Not completed — Lack of Efficacy | 1 | 1 | 5 | 0 | 7 | 9
Not completed — Physician Decision | 1 | 3 | 1 | 3 | 4 | 1
Not completed — Adverse Event | 2 | 1 | 3 | 1 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 3 | 0 | 3 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other than specified above | 0 | 2 | 11 | 3 | 5 | 3

BASELINE CHARACTERISTICS:
Population: Baseline population included safety analysis set (SAF) that included all randomized participants who received any investigational product and analyzed as treated. One participant randomized into Dupilumab 200 mg q2w arm was not treated and hence, excluded from the baseline population.
Groups:
- Dupilumab 300 mg q2w: Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single injection of Placebo (for Dupilumab) alternating with single 300 mg injection of Dupilumab q2w from Week 1 to Week 15.
- Dupilumab 300 mg q4w: Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection of Dupilumab q4w and Placebo (for Dupilumab) qw (when Dupilumab not administered) from Week 1 to Week 15.
- Total: Total of all reporting groups
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo | Total
Number analyzed (Participants) | 63 | 64 | 61 | 65 | 65 | 61 | 379
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (10.74) | 39.4 (12.06) | 35.8 (14.90) | 36.8 (10.77) | 36.6 (11.55) | 37.2 (13.10) | 37.0 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 25 | 25 | 31 | 21 | 145
  Male | 43 | 41 | 36 | 40 | 34 | 40 | 234

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Eczema Area and Severity Index Score (EASI) From Baseline to Week 16
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Time Frame: Baseline to Week 16
Population: Full analysis set (FAS) that included all randomized participants who received at least 1 dose of study drug. Here, number of participants analyzed = participants with EASI score assessment at specified time-point. Efficacy data was set to missing after use of rescue medication. Missing values imputed by last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Deviation); unit: Percent change
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 61 | 63 | 60 | 65 | 64 | 61
Percent change | -75.5 (26.86) | -70.5 (35.09) | -67.4 (31.97) | -64.9 (37.21) | -46.7 (41.96) | -20.2 (46.15)
Statistical Analysis 1: Comparison: Dupilumab 300 mg qw vs Placebo; LS mean and standard error were obtained using analysis of covariance (ANCOVA) model with treatment and randomization strata (moderate vs severe;Japan vs rest of world) and relevant baseline values as covariates. Multiplicity was controlled using hierarchical testing procedure:highest dose vs. placebo was tested first. Comparison order was 300 mg qw,300 mg q2w,200 mg q2w,300 mg q4w & 100 mg q4w, vs placebo respectively. Testing continues only if previous comparison was statistically significant; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; Least square (LS) mean difference = -55.7, 95% CI 2-sided [-68.9 to -42.4], Standard Error of Mean 6.74 — Dupilumab 300 mg qw vs Placebo
Statistical Analysis 2: Comparison: Dupilumab 300 mg q2w vs Placebo; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -50.1, 95% CI 2-sided [-63.3 to -37.0], Standard Error of Mean 6.67 — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 3: Comparison: Dupilumab 200 mg q2w vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -47.4, 95% CI 2-sided [-60.6 to -34.1], Standard Error of Mean 6.76 — Dupilumab 200 mg q2w vs Placebo
Statistical Analysis 4: Comparison: Dupilumab 300 mg q4w vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -45.4, 95% CI 2-sided [-58.5 to -32.3], Standard Error of Mean 6.66 — Dupilumab 300 mg q4w vs Placebo
Statistical Analysis 5: Comparison: Dupilumab 100 mg q4w vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -26.8, 95% CI 2-sided [-39.8 to -13.7], Standard Error of Mean 6.65 — Dupilumab 100 mg q4w vs Placebo

2. Secondary Outcome: Percentage of Participants Who Achieved Investigator's Global Assessment (IGA) Response at Week 16
Description: IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a static 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear). Values after first rescue medication were set to missing and participants with missing IGA score at Week 16 were treated as a non-responders.
Time Frame: Week 16
Population: Analysis was performed on FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 63 | 64 | 61 | 65 | 65 | 61
Percentage of participants | 33.3 [21.95 to 46.34] | 29.7 [18.91 to 42.42] | 27.9 [17.15 to 40.83] | 21.5 [12.31 to 33.49] | 12.3 [5.47 to 22.82] | 1.6 [0.04 to 8.80]

3. Secondary Outcome: Percentage of Participants Who Achieved IGA Score Reduction of ≥2 at Week 16
Description: IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic success is an IGA score of 0 (clear) or 1 (almost clear). Participants with IGA score reduction from baseline of ≥2 points at Week 16 were reported. Values after first rescue medication were set to missing and participants with missing IGA score at Week 16 were treated as a non-responders.
Time Frame: Week 16
Population: Analysis was performed on FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 63 | 64 | 61 | 65 | 65 | 61
Percentage of participants | 50.8 [37.89 to 63.62] | 46.9 [34.28 to 59.77] | 42.6 [30.04 to 55.94] | 35.4 [23.92 to 48.23] | 20.0 [11.10 to 31.77] | 9.8 [3.70 to 20.19]

4. Secondary Outcome: Percent Change in Peak Weekly Averaged Pruritus Numerical Rating Scores (NRS) From Baseline to Week 16
Description: Pruritus NRS is an assessment tool that is used to report the intensity of participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]).
Time Frame: Baseline to Week 16
Population: Analysis was performed on FAS. Here, number of participants analyzed = participants with pruritus NRS assessment at specified time-point. Efficacy data was set to missing after use of rescue medication. Missing values imputed by LOCF.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 62 | 63 | 58 | 63 | 64 | 58
Percent change | -52.85 (31.368) | -46.22 (31.964) | -40.6 (33.073) | -38.69 (38.366) | -21.47 (32.952) | -0.43 (38.423)

5. Secondary Outcome: Absolute Change in Peak Weekly Averaged Pruritus NRS From Baseline to Week 16
Description: as for outcome 4
Time Frame: Baseline to Week 16
Population: Analysis was performed on FAS. Here, number of participants analyzed =participants with pruritus NRS assessment at specified time-points. Efficacy data was set to missing after use of rescue medication. Missing values imputed by LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 63 | 64 | 61 | 65 | 65 | 61
units on a scale
  Baseline: number analyzed (Participants) | 62 | 63 | 59 | 63 | 64 | 58
  Baseline | 6.54 (1.54) | 6.74 (2.072) | 6.98 (2.315) | 6.84 (1.853) | 6.71 (1.882) | 6.34 (1.832)
  Week 16: number analyzed (Participants) | 63 | 64 | 61 | 64 | 65 | 61
  Week 16 | 3.07 (2.148) | 3.64 (2.388) | 4.21 (2.763) | 3.99 (2.449) | 5.26 (2.465) | 6.05 (2.312)
  Change at Week 16: number analyzed (Participants) | 62 | 63 | 59 | 63 | 64 | 58
  Change at Week 16 | -3.48 (2.32) | -3.16 (2.467) | -2.77 (2.595) | -2.79 (2.609) | -1.46 (2.038) | -0.27 (2.28)

6. Secondary Outcome: Absolute Change in EASI Score From Baseline to Week 16
Description: as for outcome 1
Time Frame: Baseline to Week 16
Population: Analysis was performed on FAS. Here, number of participants analyzed = participants with EASI score assessment at specified time-points. Efficacy data was set to missing after use of rescue medication. Missing values imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 63 | 64 | 61 | 65 | 65 | 61
Units on a scale
  Baseline | 30.1 (11.23) | 33.8 (14.52) | 32.9 (15.5) | 29.4 (11.48) | 32.2 (13.49) | 32.9 (13.77)
  Week 16: number analyzed (Participants) | 61 | 63 | 60 | 65 | 64 | 61
  Week 16 | 7.2 (8.83) | 10.7 (12.89) | 10.9 (12.41) | 9.8 (11.16) | 17.4 (15.28) | 25.6 (18.32)
  Change at Week 16: number analyzed (Participants) | 61 | 63 | 60 | 65 | 64 | 61
  Change at Week 16 | -23.1 (1.70) | -21.1 (1.68) | -20.7 (1.71) | -20.4 (1.62) | -13.8 (1.64) | -5.8 (1.71)

7. Secondary Outcome: Percent Change in SCORing Atopic Dermatitis (SCORAD) Scores From Baseline to Week 16
Description: SCORAD is a clinical tool for assessing the severity of AD developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
Time Frame: Baseline to Week 16
Population: Analysis was performed on FAS. Here, number of participants analyzed = participants with SCORAD score assessment at specified time-points. Missing values imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 61 | 63 | 60 | 65 | 64 | 60
Percent change | -56.9 (4.12) | -51.2 (4.05) | -46.0 (4.12) | -48.8 (3.95) | -26.6 (3.98) | -13.8 (4.14)

8. Secondary Outcome: Absolute Change in SCORAD Scores From Baseline to Week 16
Description: as for outcome 7
Time Frame: Baseline to Week 16
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 61 | 63 | 60 | 65 | 64 | 60
units on a scale | -38.2 (2.76) | -34.4 (2.71) | -30.9 (2.76) | -33.1 (2.64) | -18.0 (2.66) | -10.5 (2.77)

9. Secondary Outcome: Percentage of Participants Who Achieved 50%, 75% and 90% Reduction From Baseline in EASI Score (EASI-50, EASI-75 and EASI-90 Respectively) at Week 16
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-50, EASI-75 and EASI-90 responders were the participants who achieved ≥50%, ≥75% and ≥90% overall improvement in EASI score respectively from baseline to Week 16.
Time Frame: Week 16
Population: Analysis was performed on FAS. Participants with a missing EASI score at Week 16 were treated as non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 63 | 64 | 61 | 65 | 65 | 61
Percentage of participants
  Reduction of 50% | 82.5 [70.90 to 90.95] | 78.1 [66.03 to 87.49] | 62.3 [48.96 to 74.39] | 70.8 [58.17 to 81.40] | 44.6 [32.27 to 57.47] | 29.5 [18.52 to 42.57]
  Reduction of 75% | 60.3 [47.20 to 72.43] | 53.1 [40.23 to 65.72] | 55.7 [42.45 to 68.45] | 49.2 [36.60 to 61.93] | 29.2 [18.60 to 41.83] | 11.5 [4.74 to 22.22]
  Reduction of 90% | 36.5 [24.73 to 49.60] | 29.7 [18.91 to 42.42] | 31.1 [19.90 to 44.29] | 29.2 [18.60 to 41.83] | 15.4 [7.63 to 26.48] | 3.3 [0.40 to 11.35]

10. Secondary Outcome: Percentage of Participants Who Achieved 50%, 75% and 90% Reduction From Baseline in SCORAD Score (SCORAD-50, SCORAD-75 and SCORAD-90 Respectively) at Week 16
Description: SCORAD is a clinical tool for assessing the severity of AD developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease). SCORAD-50, SCORAD-75 and SCORAD-90 responders were the participants who achieved ≥50%, ≥75% and ≥90% overall improvement in SCORAD score respectively from baseline to Week 16.
Time Frame: Week 16
Population: Analysis was performed on FAS. Participants with a missing SCORAD score at Week 16 were treated as non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 63 | 64 | 61 | 65 | 65 | 61
Percentage of participants
  Reduction of 50% | 68.3 [55.3 to 79.4] | 59.4 [46.4 to 71.5] | 52.5 [39.3 to 65.4] | 55.4 [42.5 to 67.7] | 26.2 [16.0 to 38.5] | 19.7 [10.6 to 31.8]
  Reduction of 75% | 23.8 [14.0 to 36.2] | 25.0 [15.0 to 37.4] | 16.4 [8.2 to 28.1] | 21.5 [12.3 to 33.5] | 7.7 [2.5 to 17.0] | 3.3 [0.4 to 11.3]
  Reduction of 90% | 6.3 [1.8 to 15.5] | 6.3 [1.7 to 15.2] | 4.9 [1.0 to 13.7] | 3.1 [0.4 to 10.7] | 3.1 [0.4 to 10.7] | 0.0 [0.0 to 5.9]

11. Secondary Outcome: Percent Change in Patient Oriented Eczema Measure (POEM) Scores From Baseline to Week 16
Description: POEM is a 7-item questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]).
Time Frame: Baseline to Week 16
Population: Analysis was performed on FAS. Here, number of participants analyzed = participants with POEM score assessment at specified time-points. Missing values imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 61 | 63 | 59 | 65 | 64 | 59
Percent change | -57.3 (4.52) | -44.0 (4.44) | -49.2 (5.54) | -46.6 (4.33) | -14.2 (4.35) | 0.2 (4.61)

12. Secondary Outcome: Absolute Change in POEM Scores From Baseline to Week 16
Description: as for outcome 11
Time Frame: Baseline to Week 16
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 61 | 63 | 59 | 65 | 64 | 59
units on a scale | -12.1 (0.88) | -9.8 (0.87) | -10.4 (0.89) | -9.9 (0.85) | -3.3 (0.85) | -1.1 (0.90)

13. Secondary Outcome: Changes in Global Individual Signs Score (GISS) Components (Erythema, Infiltration/Papulation, Excoriations, and Lichenification) From Baseline to Week 16
Description: Individual components of the AD lesions (erythema, infiltration/papulation, excoriations, and lichenification) were rated globally (each assessed for the whole body, not by anatomical region) on a 4-point scale (0=none, 1=mild, 2=moderate and 3=severe) using the EASI severity grading criteria. Total score ranges from 0 (absent disease) to 12 (severe disease).
Time Frame: Baseline to Week 16
Population: Analysis was performed on FAS. Here, number of participants analyzed = participants with GISS score assessment at specified time-points. Missing values imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 61 | 63 | 60 | 65 | 64 | 61
units on a scale
  Erythema | -0.9 (0.10) | -0.9 (0.10) | -0.8 (0.10) | -0.8 (0.10) | -0.4 (0.10) | -0.2 (0.10)
  Infiltration/Papulation | -1.2 (0.11) | -1.1 (0.11) | -1.0 (0.11) | -1.1 (0.10) | -0.6 (0.11) | -0.3 (0.11)
  Excoriations | -1.4 (0.11) | -1.4 (0.11) | -1.1 (0.11) | -1.3 (0.11) | -0.6 (0.11) | -0.4 (0.11)
  Lichenification | -1.1 (0.12) | -1.1 (0.11) | -1.0 (0.12) | -1.1 (0.11) | -0.7 (0.11) | -0.3 (0.12)

14. Secondary Outcome: Changes in GISS Cumulative Score From Baseline to Week 16
Description: Individual components of the AD lesions (erythema, infiltration/papulation, excoriations, and lichenification) were rated globally (each assessed for the whole body, not by anatomical region) on a 4-point scale (0 = none,1 = mild, 2 = moderate and 3 = severe) using the EASI severity grading criteria. Total score ranges from 0 (absent disease) to 12 (severe disease).
Time Frame: Baseline to Week 16
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Number analyzed (Participants) | 61 | 63 | 60 | 65 | 64 | 61
units on a scale | -4.6 (0.38) | -4.5 (0.37) | -3.9 (0.38) | -4.3 (0.37) | -2.3 (0.37) | -1.2 (0.38)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Baseline to Week 32) regardless of seriousness or relationship to investigational product
Description: TEAEs that developed during the treatment and follow-up period (time period from the administration of first dose of study drug to the EOS visit [Week 32]).
Groups:
- Dupilumab 300 mg qw: Participants who received 2 subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection qw from Week 1 to Week 15.
- Dupilumab 300 mg q2w: Participants who received 2 subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single injection of Placebo (for Dupilumab) alternating with single 300 mg injection of Dupilumab q2w from Week 1 to Week 15.
- Dupilumab 200 mg q2w: Participants who received 2 subcutaneous injections of Dupilumab 200 mg (for a total of 400 mg) as a loading dose on Day 1, followed by a single injection of Placebo (for Dupilumab) alternating with single 200 mg injection of Dupilumab q2w from Week 1 to Week 15.
- Dupilumab 300 mg q4w: Participants who received 2 subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection of Dupilumab q4w and Placebo (for Dupilumab) qw when Dupilumab not administered from Week 1 to Week 15.
- Dupilumab 100 mg q4w: Participants who received 2 subcutaneous injections of Dupilumab 200 mg (for a total of 400 mg) as a loading dose on Day 1, followed by a single 100 mg injection of Dupilumab q4w and Placebo (for Dupilumab) qw when Dupilumab not administered from Week 1 to Week 15.
- Placebo: Participants who received 2 subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1 followed by a single injection every week (qw) from Week 1 to Week 15.
Arm/Group | Dupilumab 300 mg qw | Dupilumab 300 mg q2w | Dupilumab 200 mg q2w | Dupilumab 300 mg q4w | Dupilumab 100 mg q4w | Placebo
Serious Adverse Events (participants affected / at risk) | 1/63 | 2/64 | 1/61 | 3/65 | 5/65 | 4/61
Other Adverse Events (participants affected / at risk) | 35/63 | 34/64 | 34/61 | 39/65 | 38/65 | 38/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 300 mg qw (N=63) | Dupilumab 300 mg q2w (N=64) | Dupilumab 200 mg q2w (N=61) | Dupilumab 300 mg q4w (N=65) | Dupilumab 100 mg q4w (N=65) | Placebo (N=61)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 300 mg qw (N=63) | Dupilumab 300 mg q2w (N=64) | Dupilumab 200 mg q2w (N=61) | Dupilumab 300 mg q4w (N=65) | Dupilumab 100 mg q4w (N=65) | Placebo (N=61)
Conjunctivitis (Eye disorders) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 3 (5) | 2 (4) | 6 (9) | 3 (3) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 3 (3)
Herpes simplex (Infections and infestations) | 1 (1) | 2 (2) | 3 (4) | 1 (1) | 5 (7) | 0 (0)
Nasopharyngitis (Infections and infestations) | 16 (23) | 16 (18) | 16 (25) | 21 (29) | 20 (29) | 16 (23)
Oral herpes (Infections and infestations) | 0 (0) | 3 (5) | 2 (4) | 3 (4) | 5 (8) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 6 (8) | 2 (2) | 5 (6) | 5 (7) | 11 (11)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (5) | 6 (7) | 3 (3) | 2 (2) | 2 (2)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 4 (5) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (16) | 2 (3) | 0 (0) | 2 (5) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 8 (40) | 5 (13) | 9 (24) | 5 (6) | 7 (18) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 8 (9) | 13 (19) | 8 (10) | 10 (12) | 11 (13) | 10 (12)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.